CLINICAL TRIAL: NCT07317284
Title: Evaluation of Peripheral Neurological Integrity and Synergistic Treatment of Photobiomodulation and Therapy Ultrasound in Patirnts With Diabetes Mellitus (Type II): Clinical Study
Brief Title: Evaluation and Treatment for Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Juliana da Silva Amaral Bruno, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: JSAmaralBruno
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Neuropathy Peripheral
Keywords: Diabetes Mellitus 2 Type; Diabetic Neuropathy; Photobiomodulation Therapy; Ultrasound Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: The clinical trial was randomized, with 60 volunteers (men and women) with diabetes mellitus (type II) following the inclusion and exclusion criteria. To form the experimental groups, three pots (1, 2, 3) were prepared, and the distribution of participants into the groups respected the degree of neuropathic impairment, classified as mild (pot 1), moderate (pot 2), or severe (pot 3) based on the results obtained by assessing nerve conduction velocity measured by the DPN Check® equipment, then used to assess sural nerve function. Sixty envelopes, numbered sequentially from 1 to 60, were also prepared and placed in the jars, using simple randomization. Even numbers were assigned to Group 1, which received synergistic treatment with photobiomodulation and therapeutic ultrasound; and odd numbers were assigned to Group 2, which received sham treatment (control group). Thus, each participant was instructed to choose an envelope from the jar corresponding to their level of impairment, in order
Who Masked: Participant, Investigator
Masking Description: The study's methodological design was double-blind: the evaluators responsible for measuring the outcomes had no prior knowledge of the type of intervention the participants underwent; and the participants themselves were also unaware of which treatment (active or sham) they were receiving. It is worth noting that the researchers responsible for administering the intervention were unaware of the results of the participants' initial assessments and did not participate in the final analyses. This methodological structure directly contributed to reducing observational and analytical biases, promoting greater reliability of the findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic Peripheral Neuropathy in Early Stages: Photobiomodulation and Therapeutic Ultrasound Treatm (Active Comparator): Arm experimental:
  Participants allocated to the experimental arm will receive a combined photobiomodulation (PBM) and therapeutic ultrasound (TUS) protocol applied bilaterally over the anatomical pathway of the sural nerve. TUS parameters: 1 MHz frequency, pulsed mode (50% duty cycle), secondary frequency of 100 Hz, intensity of 0.8 W/cm², energy density of 144 J/cm². PBM parameters: 808-nm infrared wavelength, continuous mode, 100 mW power, irradiation area of 0.125 cm², resulting in 36 J total energy per session (286 J/cm²).
  Interventions: Device: Active Comparator
- Early diabetic peripheral neuropathy: Sham Group (Sham Comparator): Arm Control (Sham):
  Participants allocated to the control arm will undergo a sham procedure designed to mimic the experimental intervention without delivering therapeutic energy. The same device will be used with minimal TUS settings: 1 MHz frequency, 50% duty cycle, secondary frequency of 16 Hz, intensity of 0.1 W/cm², energy density of 18 J/cm². The PBM emitter will remain off to ensure no light emission.
  Interventions: Device: Sham Group Arm

INTERVENTIONS:
Device: Active Comparator — Participants allocated to the experimental arm will receive a combined photobiomodulation (PBM) and therapeutic ultrasound (TUS) protocol applied bilaterally over the anatomical pathway of the sural nerve, using the Recupero device (MMOptics, São Carlos, São Paulo, Brazil), which integrates both PBM and TUS modalities for research and clinical applications.
  Therapeutic ultrasound parameters: 1 MHz frequency, pulsed mode (50% duty cycle), secondary frequency of 100 Hz, intensity of 0.8 W/cm² , energy density of 144 J/cm².
  Photobiomodulation parameters: 808-nm infrared wavelength, continuous mode, 100 mW power, irradiation area of 0.125 cm², resulting in 36 J total energy per session (286 J/cm²).
  Arms: Diabetic Peripheral Neuropathy in Early Stages: Photobiomodulation and Therapeutic Ultrasound Treatm
Device: Sham Group Arm — Participants allocated to the control arm will undergo a sham procedure designed to mimic the experimental intervention without delivering therapeutic energy. The same device will be used (RECUPERO, MMOptics, São Carlos, São Paulo, Brazil) with minimal ultrasound therapy settings: 1 MHz frequency, 50% duty cycle, secondary frequency of 16 Hz, intensity of 0.1 W/cm², energy density of 18 J/cm². The photobiomodulation emitter will remain off to ensure no light emission.
  Arms: Early diabetic peripheral neuropathy: Sham Group

SUMMARY:
This study aims:

* To compare conventional diabetic neuropathy screening techniques with user-friendly technological equipment;
* To evaluate the effects of the combined application of laser and therapeutic ultrasound in the treatment of Diabetic Peripheral Neuropathy (DPN) in its early stages, aiming to prevent severe complications, such as the development of diabetic foot.

Two groups were formed: Treatment group and placebo group. 24 sessions were performed (twice a week, on alternate days). It is concluded that the combined treatment with laser and therapeutic ultrasound for diabetic peripheral neuropathy promotes a significant reduction in symptoms and improvement in sensitivity in patients with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic disease that currently affects approximately 589 million adults, aged between 20 and 79 years, worldwide. Alarming projections indicate that, by 2050, this number could exceed 853 million individuals in the same age group. The DPN is one of the most common complications of DM, characterized by a set of syndromes with diverse clinical and subclinical manifestations. The neurological damage tends to be extensive, largely compromising the peripheral nervous system in its sensorimotor and autonomic components. The pain has variable intensity, being a constant complaint, commonly described as tingling, burning or a sensation of pins and needles in the extremities, often accompanied by abnormal sensory changes, such as allodynia and hyperalgesia. Early diagnosis of DPN and ongoing monitoring are essential, as they promote education and awareness among diabetic patients, in addition to contributing to delaying or minimizing more serious complications as the disease progresses. This study aims to compare conventional diabetic neuropathy screening techniques with technological and easy-to-use equipment and, from there, evaluate the effects of the combined application of photobiomodulation and therapeutic ultrasound in the treatment of DPN in its early stages, aiming to prevent severe complications, such as the development of diabetic foot (sensory nerve).

Sixty participants were recruited and evaluated with various DPN screening instruments. They were then randomly assigned to two groups: a treatment group and a control group.

The treatment group received combined stimulation with photobiomodulation and therapeutic ultrasound in the sural nerve region, with the following parameters: continuous laser, wavelength of 808 nm, and therapeutic ultrasound with a frequency of 1 MHz, pulsed mode, for 6 minutes on each sural nerve, with rotational movement of the transducer.

The results of objective assessments performed with the DPN Check® showed that, in the treatment group, there was an increase in the "normal" rating, while the "moderate" rating, which was predominant at baseline, increased. In subjective assessments, considering a broad analysis of nerve fiber types, the "normal" rating increased while the "moderate" rating decreased. In the control group, the "normal" rating remained low, and the "moderate" rating remained at 70% in objective assessments. In the subjective evaluations, there was no change in the "normal" classification (remaining at 0% from start to finish), and the "moderate" classification varied little.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes diagnosed between 7 and 15 years old;
* Age between 45 and 70 years;
* Sex female and male.

Exclusion Criteria:

* Diabetic foot;
* Lower limb involvement with metal implants, ankle and foot fractures;
* Serious illnesses such as malignant or benign tumors;
* Serious psychological problems;
* Hormonal disorders;
* Pacemaker users;
* Hemodialysis treatment;
* Drug use;
* Physiotherapy treatment for less than six months.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change in neuropathic pain intensity | Baseline and after 12 weeks of intervention.
  Changes in the severity of neuropathic symptoms (pain, burning, tingling, and numbness) in patients with diabetic peripheral neuropathy were evaluated using the following instruments: (1) Neuropathy Disability Score (NDS), a clinical scale that quantifies neuropathic severity through neurological examination. Scores range from 0 to 10 points, with higher values indicating greater neurological impairment and worse clinical outcomes, and lower values reflecting better neurological function. (2) DPN-Check, a validated point-of-care diagnostic device used to assess diabetic peripheral neuropathy by measuring sural nerve conduction velocity (NCV, m/s) and sensory nerve action potential (SNAP) amplitude (µV) through a standardized, noninvasive electrophysiological assessment. The device reports NCV values from 20 to 70 m/s and SNAP amplitude values from 0 to 32 µV. Values ≥ 4 µV and ≥ 40 m/s are considered normal, whereas lower values indicate peripheral nerve dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Vanderlei Bagnato, Phd, Study Director — University São Paulo; Cleber Ferraresi, Phd, Study Chair — University Federal of São Carlos
Locations (1):
- Research, Innovation and Development Support Center, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang J, Wu Y, Li J, et al. Synergistic effects of photobiomodulation and mechanical stimulation on nerve regeneration. Lasers in Medical Science. 2022;37(4):1931-1942. PMID: 35184274
- [Result] Paolillo FR, Paolillo AR, Joao JP, Frasca D, Duchene M, Joao HA, Bagnato VS. Ultrasound plus low-level laser therapy for knee osteoarthritis rehabilitation: a randomized, placebo-controlled trial. Rheumatol Int. 2018 May;38(5):785-793. doi: 10.1007/s00296-018-4000-x. Epub 2018 Feb 26. PMID 29480363
- [Result] Cheng K, Martin LF, Slepian MJ, Patwardhan AM, Ibrahim MM. Mechanisms and Pathways of Pain Photobiomodulation: A Narrative Review. J Pain. 2021 Jul;22(7):763-777. doi: 10.1016/j.jpain.2021.02.005. Epub 2021 Feb 23. PMID 33636371
- See also: Description Optics and Photonics Research Center — http://cepof.ifsc.usp.br/